CLINICAL TRIAL: NCT05386576
Title: Venetoclax in Combination With Asparaginase-Containing Pediatric-Inspired Chemotherapy in Adult Patients With Newly Diagnosed Acute Lymphoblastic Leukemia
Brief Title: A Study of Venetoclax in Combination With Chemotherapy to Treat Newly Diagnosed Acute Lymphoblastic Leukemia (ALL)
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-372
Record Dates: First submitted 2022-05-18; First posted 2022-05-23 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Venetoclax; 21-372
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — venetoclax

STUDY DESIGN:
Intervention Model Description: This is a phase I single-arm, single-center study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Venetoclax in Combination With Chemotherapy (Experimental): All patients will complete Induction I and II of the treatment regimens, consisting of several chemotherapy agents including Peg-ASP.
  Interventions: Drug: Venetoclax

INTERVENTIONS:
Drug: Venetoclax — During Induction I, for patients on Dose Level 1, venetoclax will be administered at a dose of 100mg on day 5, 200mg on day 6 and 400mg on days 7-28. For patients on Dose Level 01, venetoclax will be administered at a dose of 100mg on day 5 and 200mg on days 6-28.
  During Induction II, venetoclax will be administered at either 400mg daily (Dose Level 1) or 200mg daily (Dose Level -1) from days 1-14 and 29-42.

SUMMARY:
The researchers are doing this study to find out whether combining venetoclax with several different standard chemotherapy drugs used to treat acute lymphoblastic leukemia (ALL) in children is safe and effective in adults with newly diagnosed ALL. Participants in this study will be under the age of 60, and they will have T- or B-cell ALL.

DETAILED DESCRIPTION:
All patients will complete Induction I and II of the treatment regimens, consisting of several chemotherapy agents including Peg-ASP.

* For Dose Level 1: Venetoclax will be administered at a dose of 100mg on day 5, 200mg on day 6 and 400mg on days 7-28 during Induction I. During Induction II, venetoclax will be administered at 400mg daily from days 1-14 and 29-42.
* For Dose Level -1: Venetoclax will be administered at a dose of 100mg on day 5 and 200mg on days 6-28 during Induction I. During Induction II, venetoclax will be administered at 200mg daily from days 1-14 and 29-42.
* Bone marrow aspirate and biopsy will be performed at day 14 of Induction I, after Induction I and Induction II for disease assessment.

For those who remain on study after Induction II, they will proceed to consolidation therapy. Consolidation blocks contain 2 Intensification blocks (22 days each) and 2 Re-Induction blocks (43 days each), consisting of several chemotherapy agents including Peg-ASP.

* Venetoclax will be administered at a dose of 400mg daily (Dose Level 1) or 200mg daily (Dose Level -1) from days 1-22 during Intensification blocks, and from days 1-14 and 29-42 during Re-Induction blocks.
* Bone marrow aspirate and biopsy will be performed after Re-Induction I and Re-Induction II for disease assessment.
* Patients who relapse either with MRD or morphologically will be removed from study to pursue alternative therapy.
* Patients who remain in MRD negative CR will remain on study and proceed to Maintenance.
* Maintenance block contains 4-drug regimen (vincristine, oral methotrexate, oral mercaptopurine, and prednisone) for 2 years. No venetoclax will be administered during this block. Bone marrow aspirate and biopsy will be performed every 3 months during the Maintenance block. Patients who remain in MRD negative CR will remain on study to complete the study treatment. Patients who relapse either with MRD or morphologically will be removed from study to pursue alternative therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with newly diagnosed Philadelphia chromosome (Ph) negative ALL.
* Patients with T- or B-cell lymphoblastic lymphoma with no bone marrow involvement will also be eligible for the study.
* Age 18-60
* ECOG performance status of 0-2
* Adequate renal function as demonstrated by a calculated creatinine clearance of ≥ 60 ml/min.
* Adequate hepatic function as demonstrated by a total bilirubin ≤ 2.0 mg/dl (unless attributable to Gilbert's disease) and an alkaline phosphatase, AST, and ALT ≤ 4 times the upper limit of normal (unless clinically considered to be related to liver involvement with leukemia)
* Patients with central nervous system (CNS) involvement by ALL are eligible and may receive concomitant treatment with radiation therapy and/or intrathecal chemotherapy in accordance with standard medical practice. For patients with CNS disease, dexamethasone may be temporarily administered instead of prednisone to reduce CNS pressure, at the discretion of the treating physician and after discussion with the MSK PI. Once dexamethasone is no longer needed, prednisone should be given as per protocol for 28 days.
* Negative serum pregnancy test in women of childbearing potential

Exclusion Criteria:

* CML in lymphoid blast crisis, mature B-cell (i.e. Burkitt's) lymphoma or mixed phenotype acute leukemia (MPAL)
* Prior treatments for ALL, except any doses of corticosteroids and hydroxyurea or one dose of vincristine
* Patients who received strong and/or moderate CYP3A inducers within 7 days prior to the initiation of study treatment
* Unstable angina and/or MI or stroke within 6 months prior to screening, and/or impaired cardiac function with EF <40% or NYHA class III/IV
* Pregnant or lactating women. Women and men of childbearing age should use effective contraception while on this study and continue for 1 year after all treatment is finished.
* Patients with HIV or active hepatitis B or hepatitis C infection are ineligible.
* Patients with concurrent active malignancies as defined by malignancies requiring any therapy other than expectant observation or hormonal therapy, with the exception of squamous and basal cell carcinoma of the skin, in situ cervical cancer, adequately treated stage I/II cancer from which the patient is current in complete remission, or any other cancer from which the patient has been disease free for five years.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-06-16 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
proportion of patients who have a Dose Limiting Toxicities | up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jae Park, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm